CLINICAL TRIAL: NCT06766708
Title: The Effect of a Self-Management Lymphedema Education Program on Lymphedema, Lymphedema-Related Symptoms, Patient Compliance, Daily Living Activities and Patient Activation in Patients With Breast Cancer-Related Lymphedema: A Quasi-Experimental Study
Brief Title: The Effect of a Self-Management Lymphedema Education Program on Lymphedema, Symptoms, Compliance, Daily Living Activities, and Patient Activation in Breast Cancer-Related Lymphedema: A Quasi-Experimental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gizem Cansiz Ucar (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Sponsor-Investigator, Gizem Cansiz Ucar, Principal Investigator, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KA-19098
Record Dates: First submitted 2024-12-17; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer Survivor; Lymphedema
Keywords: Breast cancer-related lymphedema; daily life activities; patient activation; patient adaptation; patient education; self-management of lymphedema
MeSH Terms: conditions — Lymphedema; Breast Cancer Lymphedema; Patient Participation

STUDY DESIGN:
Intervention Model Description: this pre-test post-test in one group quasi-experimental study
Masking Description: In our study, single-blinded research was implemented by blinding the researcher. Bilateral upper extremity circumferences of the patients were measured at 10 different points, spaced 4 cm apart from the wrist to the axilla, by an expert nurse other than the researcher. The measurements were recorded with an accuracy of up to 0.1 cm.
  During the initial interview with the patients, the researcher completed the scales and forms and then conducted the Lymphedema Management Education Program using an educational booklet developed by the researchers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental grup (Experimental): one group quasi-experimental study was to determine the effects of self-management lymphedema (SML) education program on the patient adherence, daily life activities and patient activation in patients with breast- cancer related lymphedema (BCRL).
  Interventions: Other: self-management lymphedema (SML) education program

INTERVENTIONS:
Other: self-management lymphedema (SML) education program — The content of the booklet was prepared based on literature review.. In addition to the above intervention methods, the phone number of each patient was taken and the patients were followed up by phone for 12 months. For this purpose, the patient was asked to fill in the compliance chart prepared in order to monitor the patient's compliance and was checked by the researcher every two weeks by phone call. By phone call; compliance with skin care, SLD, compression garments and exercise practices included in the SMLEP were evaluated and recorded. Within the scope of the SMLEP, the patients were asked to do exercises and SLD at least 3 days a week and 2 times a day (morning and evening) for 12 months. It was recommended to wear compression garments, especially during exercises and throughout the day.

SUMMARY:
The aim of this pre-test post-test quasi-experimental study is to evaluate the effects of a self-management lymphedema (SML) education program on patient adherence, daily life activities, and patient activation in individuals with breast cancer-related lymphedema (BCRL). This study involves 44 patients diagnosed with BCRL and is conducted at Hacettepe University Oncology Hospital Lymphedema Diagnosis and Treatment Application and Research Center. Upper extremity lymphedema assessments are performed at the beginning of the study, followed by the implementation of a structured SML education program. Participants are monitored for a total of 12 months. Data collection tools include the Personal Information Form, Upper Extremity Lymphedema Diagnosis Form, Adaptation to Chronic Illness Scale, KATZ Daily Living Activities Index, Disability of Arm, Shoulder, and Hand Questionnaire, and Patient Activation Measure.

DETAILED DESCRIPTION:
This study focuses on evaluating the potential benefits of a structured self-management lymphedema education program in patients with breast cancer-related lymphedema. It aims to improve patient adherence, activation, and daily life activity levels through a comprehensive education-based intervention.The study was conducted as a master's thesis and has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Being female,
* Aged 18 years or older,
* Having undergone axillary lymph node dissection,
* Having undergone breast cancer surgery,
* Diagnosed with lymphedema (stage 1-2),
* Individuals with no surgical plans during the study period.

Exclusion Criteria:

* Not diagnosed with lymphedema,
* Having a medical condition that prevents exercise,
* Having advanced-stage heart or kidney failure,
* Patients who refused to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since individuals diagnosed with breast cancer are predominantly women, the sample consisted of female participants.
Enrollment: 44 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
The Impact of a Lymphedema Management Education Program on Symptoms in Breast Cancer-Related Lymphedema Patients Using Circumferential Measurements and Bioimpedance Spectroscopy (BIS) | By the end of the program (after 12 months).
  The impact of the Lymphedema Management Education Program will be evaluated on symptoms in breast cancer-related lymphedema patients using circumferential measurements and bioimpedance spectroscopy (BIS). Measurements will involve taking circumferential readings at 4 cm intervals along the arm with a 1-inch retractable tape, and arm volumes will be calculated using the truncated cone formula. BIS will provide L-Dex ratios to identify subclinical (≥6.5) and clinical (≥7) lymphedema through the L-Dex U400® device. Lymphedema severity will be classified based on the Tracey-Volume and Stilwell systems by comparing volume differences between affected and unaffected limbs. Baseline and endpoint measurements will be conducted under standardized conditions by a specialist nurse to ensure accuracy and consistency.
The Impact of a Lymphedema Management Education Program on Patient Compliance Using the Patient Activation Measure (PAM) | By the end of the program (after 12 months)
  The impact of the Lymphedema Management Education Program on patient compliance will be evaluated using the Patient Activation Measure (PAM).
The Impact of a Lymphedema Management Education Program on Activity Levels Using the Patient Activation Measure (PAM) | By the end of the program (after 12 months).
  The impact of the Lymphedema Management Education Program on activity levels will be evaluated using the Patient Activation Measure (PAM)
The Impact of a Lymphedema Management Education Program on Activity Levels Using the Daily Living (Katz ADL) Index | By the end of the program (after 12 months).
  The impact of the Lymphedema Management Education Program on activity levels will be evaluated using the Katz Activities of Daily Living (Katz ADL) Index.
The Impact of a Lymphedema Management Education Program on Independence in Daily Living Activities Using the Katz Activities of Daily Living (Katz ADL) Index | By the end of the program (after 12 months).
  The measurement of independence in daily tasks (e.g., bathing, dressing) will be conducted using the Katz Activities of Daily Living (Katz ADL) Index.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cansiz G, Arikan Donmez A, Kapucu S, Borman P. The effect of a self-management lymphedema education program on lymphedema, lymphedema-related symptoms, patient compliance, daily living activities and patient activation in patients with breast cancer-related lymphedema: A quasi-experimental study. Eur J Oncol Nurs. 2022 Feb;56:102081. doi: 10.1016/j.ejon.2021.102081. Epub 2021 Dec 1. PMID 34875398
- See also: Related Info — https://doi.org/10.1016/j.ejon.2021.102081